CLINICAL TRIAL: NCT00754676
Title: Randomized Single Blind Trial of Endoscopic Stenting for Chronic Pancreatitis-Associated Abdominal Pain
Brief Title: Endoscopic Stenting for Chronic Abdominal Pain
Status: Completed | Type: Observational
Sponsor: Leigh Powell (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Alabama at Birmingham (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Leigh Powell, Principle Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Other Study IDs: F040924005; 5K24DK070629-05 (NIH)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The prospective sham randomized study will evaluate the role of endoscopic stenting inpatients with chronic pancreatitis and chronic abdominal pain.

DETAILED DESCRIPTION:
Endoscopic stenting is increasingly used for the treatment of a variety of pancreatic disorders. Although a number of studies suggest that pancreatic stenting relieves abdominal pain in approximately 70% of patients, there has been no randomized study. Since any intervention may improve pain, the effectiveness of endoscopy cannot be ascertained without a true placebo arm or sham therapy group.

The study will aim to determine the effectiveness of pancreatic stents in relieving chronic pain in the setting of chronic pancreatitis. Since these procedures do carry risk, a placebo controlled fashion is used for this study

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to the principal investigator for chronic pancreatitis will be enrolled.

Exclusion Criteria:

* There are no gender nor racial exclusion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women diagnosed with chronic pancreatitis.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2004-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Wilcox, M.D., Principal Investigator — University of Alabama at Birmingham